CLINICAL TRIAL: NCT04076345
Title: Interest of the Presepsin Assay as a Biomarker of Bacterial Infection, in the Management of Newborns and Infants Under 3 Months of Age Admitted for Fever in Pediatric Emergency Service
Brief Title: Interest of the Presepsin Assay as a Biomarker of Bacterial Infection, in the Management of Newborns and Infants Under 3 Months of Age Admitted for Fever in Pediatric Emergency Service (Presepsin)
Acronym: presepsin
Status: Terminated | Type: Observational
Why Stopped: investigator not available
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Mitsubishi Chemical Europe (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 POIRIER; 2019-A00704-53 (Other: ANSM)
Record Dates: First submitted 2019-08-26; First posted 2019-09-03 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Newborn Sepsis; Fever
Keywords: presepsin; biomarker; newborns; infants under 3 months of age; fever; paediatric emergency
MeSH Terms: conditions — Neonatal Sepsis; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bacterial group: Newborns or infants less dans 3 months old with fever and positive bacterial sample.
  Interventions: Diagnostic Test: Prespesin assay on PATHFAST analyser
- Viral group: Newborns or infants less dans 3 months old with fever and positive viral sample.
  Interventions: Diagnostic Test: Prespesin assay on PATHFAST analyser
- Negatives Microbiological samples: Newborns or infants less dans 3 months old with fever and negatives microbiological samples.
  Interventions: Diagnostic Test: Prespesin assay on PATHFAST analyser

INTERVENTIONS:
Diagnostic Test: Prespesin assay on PATHFAST analyser — Collection of parental non-opposition by the doctor taking care of the child. Addition of an additional 500μl tube to the usual blood sampling as part of the protocol for the management of children under 3 months of age with fever. This blood test contains CRP, PCT, NFS, Hemoculture.
  There is no additional venipuncture. This blood sample is taken by the nurse after parental non-opposition. Transfer of the sample to the laboratory. In the laboratory, centrifugation of the sample, taking the plasma alone which will be frozen.
  Delayed assay of presepsin, in series, after thawing of samples. Collection of data and analyzes by the principal investigator in collaboration with the statistician methodologist.
  The immunoassay of presepsin with PATHFAST is based on chemiluminescence.

SUMMARY:
The purpose of this study is to validate presepsin as a biological marker for identifying bacterial fever among febrile syndromes of infants under three months of age. Clearly, our goal is to determine if this marker can help us distinguish a viral infection from a bacterial infection. Indeed, presepsin would be specific for bacterial infection, and rise earlier in the blood during infection than biological markers currently used. Such validation could improve the precocity of the therapeutic management by a better targeted antibiotic therapy, and the limitation of invasive complementary examinations (lumbar puncture), in infants for whom the fear of a bacterial infection leads to examinations and systematic treatments.

DETAILED DESCRIPTION:
An exploratory proof of concept that evaluates an innovative and minimally invasive diagnostic technique, with brief, monocentric longitudinal follow-up, this study aims to validate presepsin as a biomarker for identifying bacterial fever among febrile syndromes of infants under three months of age. Presepsin is thought to be specific for sepsis, and would rise earlier in the blood during sepsis than biomarkers currently used. Such validation could improve the precocity of the therapeutic management by a better targeted antibiotic therapy, and the limitation of invasive complementary examinations (lumbar puncture), in infants for whom the fear of a bacterial infection leads to examinations and systematic treatments.

To do this, we will study the discriminative power (bacterial or viral, verified, a posteriori, by the results of microbiological examinations such as blood cultures, cytobacteriology of urine, lumbar puncture, virological or bacteriological samples of stool and nasopharynx) and prognosis (comparison of initial signs of clinical severity and presepsin levels, length of hospitalization and hospitalization unit) of presepsin by comparing its blood levels to the usual biological markers (CRP, PCT, leukocytes, neutrophils, lymphocytes) in children less than 3 months old with fever. It will also be compared, a posteriori, the rate of presepsin between the group of children treated with antibiotics and the group of untreated children to verify that the rate of presepsin is predictive of the initiation of antibiotic treatment.

If in this study the superiority of presepsin is confirmed, it will also be evaluated, by a medico-economic study, the effect of a decision of care based on the interpretation of the blood presepsin level on downstream health costs and on the speed of care of children under 3 months with fever presenting to the emergency department by the commissioning of a delocalized analyzer. This device is, for the moment, available only in the laboratory.

The study plans to include 160 children under 3 months admitted to pediatric emergencies or pediatric resuscitation at Estaing Hospital in Clermont-Ferrand.

Participation in the study will not require additional venipuncture given the very small amount of blood sufficient for the presepsin assay. The diagnosis of the child will not be made according to the presepsin test, but according to the standard criteria, and its management will not be modified by his participation in the study. Thus, the study presents neither benefit nor risk for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Children under 3 months old with fever, a rectal temperature greater than or equal to 38 ° C, presenting at the pediatric emergency of the Estaing Hospital or directly in pediatric intensive care unit of the Estaing Hospital.
* Coverage by a social security scheme

Exclusion Criteria:

* Failure to perform a blood test
* Children who received antibiotics before admission.
* Refusal of participation by the legal representatives of the child
* Concomitant participation of the child in a therapeutic trial or other clinical study that may influence the results of this research

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 3 months old with fever, a rectal temperature greater than or equal to 38 ° C, presenting at the pediatric emergency of the Estaing Hospital or directly in pediatric intensive care unit of the Estaing Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Measure of Presepsin | Day 0
  Presepsin rate measured in picograms / milliliters, using the PATHFAST analyzer.

SECONDARY OUTCOMES:
Measure of C-reactive protein | Day 0
  CRP level in milligrams / Liter
Measure of Procalcitonin | Day 0
  PCT rate in microgram/ Liter
Length of hospital stay | through study completion, an average of one week
  comparison between the presepsin rate and the duration of hospitalization to verify the prognostic power of presepsin (Day)
Total costs | through study completion, an average of one week
  Total costs represents cost of presepsin assay, cost of CRP and PCT assay, average cost per day of a hospital stay of a febrile child less than 3 months depending on the unit, laboratory personal cost (in euros). This allows the evaluation, by a medico-economic study, of the effect of a decision of care based on the interpretation of the blood pressepsin level on the downstream health costs and on the speed of taking care of patients children under 3 months with fever presenting to the emergency department by setting up a delocalized analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: POIRIER Véronique, Principal Investigator — CHU Estaing
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Pugni L, Pietrasanta C, Milani S, Vener C, Ronchi A, Falbo M, Arghittu M, Mosca F. Presepsin (Soluble CD14 Subtype): Reference Ranges of a New Sepsis Marker in Term and Preterm Neonates. PLoS One. 2015 Dec 31;10(12):e0146020. doi: 10.1371/journal.pone.0146020. eCollection 2015. PMID 26720209
- [Background] Okamura Y, Yokoi H. Development of a point-of-care assay system for measurement of presepsin (sCD14-ST). Clin Chim Acta. 2011 Nov 20;412(23-24):2157-61. doi: 10.1016/j.cca.2011.07.024. Epub 2011 Aug 3. PMID 21839732
- [Background] Chenevier-Gobeaux C, Bardet V, Poupet H, Poyart C, Borderie D, Claessens YE. Presepsin (sCD14-ST) secretion and kinetics by peripheral blood mononuclear cells and monocytic THP-1 cell line. Ann Biol Clin (Paris). 2016 Jan-Feb;74(1):93-7. doi: 10.1684/abc.2015.1112. PMID 26743983
- [Background] Pizzolato E, Ulla M, Galluzzo C, Lucchiari M, Manetta T, Lupia E, Mengozzi G, Battista S. Role of presepsin for the evaluation of sepsis in the emergency department. Clin Chem Lab Med. 2014 Oct;52(10):1395-400. doi: 10.1515/cclm-2014-0199. PMID 24897403